CLINICAL TRIAL: NCT05472766
Title: Pilot Randomized Controlled Trial of Anticoagulation Therapy Timing in Atrial Fibrillation After Acute and Chronic Subdural Hematoma (ATTAACH)
Brief Title: Anticoagulation Therapy Timing in Atrial Fibrillation After Acute and Chronic Subdural Hematoma
Acronym: ATTAACH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to logistical challenges in conducting the trial.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3998
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2022-11

CONDITIONS: Subdural Hematoma; Atrial Fibrillation
Keywords: Direct-acting Oral Anticoagulants
MeSH Terms: conditions — Hematoma, Subdural; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early resumption of anticoagulation (Active Comparator): The standard of care DOAC at appropriate standard dose assigned by the MRP will start at day 30 +/- 7 after diagnosis of acute or chronic subdural hematoma.
  Interventions: Drug: Direct Acting Oral Anticoagulant starting at Day 30
- Delayed resumption of anticoagulation (Active Comparator): The standard of care DOAC at appropriate standard dose assigned by the MRP will start at day 90 +/- 14 after diagnosis of acute or chronic subdural hematoma.
  Interventions: Drug: Direct Acting Oral Anticoagulant starting at Day 90

INTERVENTIONS:
Drug: Direct Acting Oral Anticoagulant starting at Day 30 — Dabigatran, Rivaroxaban, Apixaban or Edoxaban at standard dose as recommended by the MRP
  Arms: Early resumption of anticoagulation
Drug: Direct Acting Oral Anticoagulant starting at Day 90 — Dabigatran, Rivaroxaban, Apixaban or Edoxaban at standard dose as recommended by the MRP
  Arms: Delayed resumption of anticoagulation

SUMMARY:
Subdural hematoma (SDH) is a common disorder that typically results from head trauma and has increased in prevalence in recent decades. Acute subdural hematomas (aSDH) are found in up to one-third of patients with severe traumatic brain injury and are associated with an unfavorable outcome in the majority of cases. Chronic subdural hematomas (cSDH) commonly occur in the elderly population which has highest risk for developing cSDH with or without minor head injuries. The combination of the aging population, higher incidence of disease in progressively older patients, and high morbidity and mortality renders SDH a growing problem within Canada with significant health-systems burden. SDH commonly recurs even after successful surgical drainage. Atrial fibrillation (AF) is one of the most common medical comorbidities in patients with cSDH, especially in the elderly, with an expected doubling of its prevalence by the year 2030. Patients with AF are at recognized risk for stroke, so anticoagulation is indicated for almost all patients. Anticoagulation is held prior to SDH drainage to minimize the risk of intraoperative and early postoperative bleeding. After surgery, the risk of SDH recurrence must be balanced against the risk of thromboembolic events such as stroke when deciding the timing of resuming anticoagulation. Currently the decision on when to restart anticoagulation after SDH is made by clinicians on an individual patient basis without any high-quality evidence to guide this decision. The two most common approaches are: 1) early resumption of anticoagulation after 30 days of diagnosis or surgery; and 2) delayed resumption of anticoagulation after 90 days of diagnosis or surgery. However, which of these approaches leads to the best functional outcomes for patients is unclear. Our pilot RCT will test the feasibility of comparing these 2 approaches in a larger multicenter RCT.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Any SDH, defined as either acute or encapsulated partially liquefied hematoma in the subdural space diagnosed on a CT scan
3. Can have surgical drainage (either burr hole or craniotomy) for aSDH and cSDH
4. On therapeutic anticoagulation (DOAC or warfarin) as standard of care therapy prior to presentation for stroke prophylaxis secondary to AF

Exclusion Criteria:

1. aSDH requiring decompressive craniectomy
2. Mechanical heart valve or moderate to severe mitral stenosis
3. Known chronic coagulopathy (elevated INR >1.5 or PTT>40s after anticoagulant reversal, thrombocytopenia with platelet count <50x109/L) that is not amenable to reversal
4. >37 days has elapsed since initial diagnosis without recruitment into the trial
5. Active gastroduodenal ulcer, urogenital or respiratory tract hemorrhage
6. Known pregnancy or breastfeeding
7. Indication for therapeutic anticoagulation other than AF
8. Pre-randomization brain CT at 2-4 weeks after initial diagnosis or surgery date reveals significant recurrence requiring surgical drainage
9. Known to be non-compliant with prior anticoagulant
10. MRP decides to restart Warfarin (as opposed to DOACs) as prophylactic anticoagulant as part of standard therapy for the patient after cSDH or aSDH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  The number of participants enrolled for each participating institution, measured as the rate of consent for patients meeting eligibility criteria in one year per institution. Reasons for non-enrollment of eligible patients will be recorded
Implementation of study protocol | Study completion ~2.5 years
  The proportion of enrolled participants who have completed follow-up measures at 90 days with complete recording of the functional outcome degree of disability

SECONDARY OUTCOMES:
Functional outcome - Degree of disability | 90 days
  Level of disability measured by the modified Rankin Scale (mRS). The mRS is a core instrument used for measuring the degree of disability or dependence in activities of daily living that is sensitive to thromboembolic and hemorrhagic complications. It is a clinician-reported measure and widely applied for evaluating stroke patient outcomes. It is a 7-level ordered categorical scale with scores ranging from 0 (no symptoms/disability) to 6 (death). The analysis will be categorized as favourable outcome (scores 0-3) versus unfavourable outcome (scores 4-6)
Functional outcome - Degree of disability | 180 days
  Level of disability measured by the modified Rankin Scale (mRS). The mRS is a core instrument used for measuring the degree of disability or dependence in activities of daily living that is sensitive to thromboembolic and hemorrhagic complications. It is a clinician-reported measure and widely applied for evaluating stroke patient outcomes. It is a 7-level ordered categorical scale with scores ranging from 0 (no symptoms/disability) to 6 (death). The analysis will be categorized as favourable outcome (scores 0-3) versus unfavourable outcome (scores 4-6)
Functional outcome - Stroke-related neurologic deficit | 90 days
  Measured using the National Institute of Health Stroke Scale (NIHSS) which is a 15-item impairment scale. It groups scores into categories based on severity, ranging from mild to very severe, with a higher score indicating a greater degree of impairment
Functional outcome - Stroke-related neurologic deficit | 180 days
  Measured using the National Institute of Health Stroke Scale (NIHSS) which is a 15-item impairment scale. It groups scores into categories based on severity, ranging from mild to very severe, with a higher score indicating a greater degree of impairment
Incidence of intracranial hemorrhage | Continuous, baseline to 180 days
  The composite outcome of clinically-important intracranial hemorrhage defined by: 1) any increase in volume of blood in the CT of at least 33%; 2) need for surgical evacuation of SDH or repeat surgical evacuation; 3) death directly related to enlarging SDH or new parenchymal bleed; 4) symptomatic bleeding in a critical non-intracranial region
Incidence of thromboembolic events | Continuous, baseline to 180 days
  Composite outcome of clinically-important thromboembolic events defined as any of: 1) symptomatic TIA; 2) symptomatic objectively-confirmed ischemic stroke; 3) symptomatic, objectively-confirmed non-CNS systemic embolism; 4) objectively proven VTE; 5) all death directly or indirectly caused by a thrombotic event

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Pirouzmand, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Mansouri A, Nassiri F, Scales D, Pirouzmand F. Anticoagulation Therapy Timing in patients with Atrial Fibrillation after Acute and Chronic Subdural Haematoma (ATTAACH): a pilot randomised controlled trial. BMJ Open. 2024 Oct 22;14(10):e090224. doi: 10.1136/bmjopen-2024-090224. PMID 39438108